CLINICAL TRIAL: NCT04566575
Title: Isthmocele - Prediction, Prevention, Diagnosis, and Management
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-01874; sp20Fellmann
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Isthmocele
Keywords: Caesarean section; Myometrium; Hydrometra; transvaginal ultrasound; Isthmocele correction
MeSH Terms: interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: trans vaginal ultrasound (TVUS) — In the TVUS, the residual myometrium is determined after surgery and the appearance of new cysts in the area of the caesarian section scar is assessed.
Other: patient questionnaire — exploratory patient questionnaire regarding satisfaction after correction of isthmocele

SUMMARY:
An Isthmocele is a scar defect or uterine niche that develops in the myometrium due to an inadequate healing process at the site of the caesarean section incision. The management of isthmocele is not standardized and a correction typically involves invasive procedures (hysteroscopy/resectoscopy, laparoscopy, vaginal surgery). This study is to investigate the effectiveness of the procedures used to treat isthmocele.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing isthmocele correction surgery within the period from 01.01.2017 to 31.12.2020 at the University Hospital Basel, Women's Hospital

Exclusion Criteria:

* Missing information on the preoperative initial situation (preoperative myometrium thickness, lack of imaging via TVUS)
* Missing information on key characteristics that are important in the collection of retrospective data analysis (e.g. data on the previous caesarean section)
* Inability to give an informed consent
* Lack of German language skills

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent surgery for isthmocele at the University Hospital Basel between 01.01.2017 and 31.12.2020. Time interval from the operation performed to the study-specific consultation has a maximum of 4 years.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Myometrium thickness after isthmocele correction procedure (mm) | single time-point at baseline (approx. 10 minutes)
  Myometrium thickness after isthmocele correction procedure (mm), compared to myometrium thickness before isthmocele correction procedure, measured by TVUS (in mm)
Occurrence of new cysts in the area of caesarean sectio after isthmocele correction procedure | single time-point at baseline (approx. 10 minutes)
  Occurrence of new cysts in the area of caesarean sectio after isthmocele correction procedure, measured by TVUS and compared to number of cysts before isthmocele correction procedure
Patient satisfaction after isthmocele correction procedure | single time-point at baseline (approx. 10 minutes)
  Patient satisfaction after isthmocele correction procedure, analysed by explorative questionnaire ( ranging from a = very satisfied to f = absolutely not satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Viola Heinzelmann, Prof. Dr. med., Principal Investigator — University Hospital Basel, Women's Hospital
Locations (1):
- University Hospital Basel, Women's Hospital, Basel, Switzerland